CLINICAL TRIAL: NCT07175883
Title: Comparison of Postoperative Pain in Primary Cemented Total Knee Arthroplasty With or Without Drain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario Reina Sofia de Cordoba (Other Government)
Responsible Party: Principal Investigator, Jesús Castellano Curado, Principal Investigator, Hospital Universitario Reina Sofia de Cordoba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HURSKNEEDRAIN
Record Dates: First submitted 2025-08-04; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Postoperative Pain; Arthropathy of Knee
Keywords: drainage; Arthroplasty, Replacement, Knee; Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Comparative prospective clinical trial between 2 groups of randomly selected patients (30 patients each)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DRAINAGE GROUP (A) (Experimental): Patients in group A will have a Redon drain placed at the end of the procedure. Both groups of patients will be explained early active flexion-extension exercises to initiate mobilization and multimodal analgesia will be provided. Patients in group A will receive perioperative care adapted to the drainage. All patients will have their baseline pain measured preoperatively and postoperatively using an analog rating scale. Patients will be checked if they require morphine rescue analgesia during their hospital stay. Postoperative pain assessment will be performed at discharge.
  Interventions: Procedure: Redon drain
- NO DRAINAGE GROUP (B) (No Intervention): Patients in group B will not have a Redon drain placed at the end of the procedure.
  Both groups of patients will be explained early active flexion-extension exercises to initiate mobilization and multimodal analgesia will be provided. All patients will have their baseline pain measured preoperatively and postoperatively using an analog rating scale. Patients will be checked if they require morphine rescue analgesia during their hospital stay. Postoperative pain assessment will be performed at discharge.

INTERVENTIONS:
Procedure: Redon drain — Patients in group A will have a Redon drain placed at the end of the procedure following the usual technique
  Arms: DRAINAGE GROUP (A)

SUMMARY:
The use of closed aspirative surgical drainage presents a truly questionable role in the field of orthopedic surgery.

The pathophysiological mechanisms on which it acts have been widely theorized, as well as the disadvantages that could be associated, both at a biological and socio-sanitary level, so that clinical guidelines opt to leave the decision to the surgeon's discretion.

Although its application and postoperative complications in knee arthroplasty are widely documented, the results are inconclusive and the scientific community does not seem to reach a consensus.

The main debate centers on bleeding during the immediate postoperative period, a classic complication of these interventions, but which seems to be being avoided with the introduction of new techniques and drugs, mainly the use of tranexamic acid.

However, a fundamental element of the postoperative period of these interventions that all the research seems to omit is pain in the postoperative period, which is key, as the pain of gonarthrosis is the main indication for the intervention.

It is because of this lack in the essential knowledge of this intervention that we propose the following hypothesis: the use of drainage in knee arthroplasty does not reduce pain during the early postoperative period.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 60 years of age
* Candidates for hybrid total knee arthroplasty with preservation of the posterior cruciate ligament

Exclusion Criteria:

* Patients with previous ipsilateral or contralateral knee surgery (contralateral knee arthroplasty, osteotomized, previous cruciate ligament or meniscal repair included)
* History of rheumatologic diseases
* History of articular infection

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-12 (Actual)

PRIMARY OUTCOMES:
Preoperative baseline pain and postoperative pain at discharge | Preoperative baseline pain (Day 0) and postoperative pain at discharge (Day 2)
  Preoperative baseline pain and postoperative pain at discharge, both assessed using an Analog Rating Scale (scale 0-10)

SECONDARY OUTCOMES:
Body Mass Index | BMI measured in Day 0 (at the time of admision in hospital)
  Weight in kilograms (kg) divided by the square of height in meters (m2)

OTHER OUTCOMES:
Use of opioid rescue during hospital stay | Measured the day of medical discharge, on average postoperative day 2
  Total opioid rescue doses administered throughout the entire period of hospitalization following surgery until medical discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Unievrsitario Reina Sofia de Córdoba, Córdoba, CORDOBA, Spain

IPD SHARING:
Plan to Share IPD: No